CLINICAL TRIAL: NCT07133698
Title: High Flow Nasal Cannula vs. High Velocity Nasal Insufflation for Weaning From Mechanical Ventilation in Respiratory ICU
Brief Title: High Flow Nasal Cannula Versus High Velocity Nasal Insufflation for Weaning
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Waleed Gamal Elddin Khaleel, Assistant professor of chest diseases, Assiut University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: WGEK-HVNI-HFNC
Record Dates: First submitted 2025-08-14; First posted 2025-08-21 (Actual); Last update posted 2025-08-21 (Actual); Status verified 2025-08

CONDITIONS: Weaning From Mechanical Ventilation
Keywords: Weaning; HFNC; HVNI; Noninvasive ventilation
MeSH Terms: interventions — Noninvasive Ventilation

STUDY DESIGN:
Intervention Model Description: Parallel Assignment: Each participant is assigned to only one of the three intervention groups (High flow nasal cannula weaning, High velocity nasal insufflation weaning, noninvasive ventilation weaning) for the entire duration of the weaning period. Outcomes are then compared between these groups.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- HFNC weaning (Experimental)
  Interventions: Device: High Flow nasal Cannula
- HVNI weaning (Experimental)
  Interventions: Device: High velocity nasal insufflation
- Noninvasive ventilation weaning (Active Comparator)
  Interventions: Device: Noninvasive ventilation

INTERVENTIONS:
Device: High Flow nasal Cannula — Eligible subjects successfully passing a SBT will be extubated and immediately randomized (1:1:1) to receive one of the following post-extubation respiratory supports for ≥24 hours:
  HVNI Arm: High-Velocity Nasal Insufflation (Flow: 40-60 L/min, FiO₂ titrated to SpO₂ ≥92%).
  Arms: HFNC weaning
Device: High velocity nasal insufflation — HFNC Arm: High-Flow Nasal Cannula (Flow: 50-60 L/min, FiO₂ titrated to SpO₂ ≥92%).
  Arms: HVNI weaning
Device: Noninvasive ventilation — NIV Arm: Non-Invasive Ventilation (Mode: [e.g., PSV], IPAP: [e.g., 8-12 cmH₂O], EPAP: [e.g., 4-6 cmH₂O], FiO₂ titrated to SpO₂ ≥92%) delivered via [e.g., oronasal mask] for ≥16 hours/day initially, with weaning per protocol.
  Arms: Noninvasive ventilation weaning

SUMMARY:
In intensive care units (ICUs), approximately 10% to 15%of patients ready to be separated from a ventilator experience extubation failure leading to reintubation. In patients considered at high risk, these rates can even exceed 20%. Because reintubation is associated with particularly high mortality a strategy of oxygenation aimed at avoiding reintubation deserves consideration. Although noninvasive ventilation may prevent postextubation respiratory failure in patients at high risk only 2 small-scale randomized clinical trials (RCTs) have shown decreased reintubation rates compared with standard oxygen. The most recent international clinical practice guidelines recommend the use of noninvasive ventilation to prevent post extubation respiratory failure in patients at high risk of extubation failure (7). However, up until now, no large-scale RCT has demonstrated a significant reduction of reintubation rates with noninvasive ventilation compared with standard oxygen. Thereby, most patients are treated with standard oxygen in clinical practice and only10% of them receive noninvasive ventilation after extubation in the ICU.

High-flow nasal cannula (HFNC) oxygen therapy is a new type of respiratory support system which can supply high flow mixed gases through special nasal prongs at a sufficient temperature and humidity for patient comfort. Many studies have confirmed that the comfort and tolerance of HFNC is significantly higher than that of NIV. As an alternative to NIV, HFNC has been shown to be as efficacious as NIV in preventing post-extubation respiratory failure or re-intubation in patients with hypoxemic respiratory failure.

High-velocity nasal insufflation, a form of high-flow nasal cannula, focuses on optimum efficiency of the dead-space purge to augment ventilation (removal of carbon dioxide from the dead space between breaths), in addition to providing other effects of high-flow nasal cannula. This is accomplished by use of small-bore nasal cannulae (typically 2.7-mm internal diameter for adult patients) to produce high velocity flow that is approximately 360% greater than that of the larger bore cannulae used in previous studies. According to flow analyses8 and clinical experience, high velocity nasal insufflation typically requires a flow of 25 to 35 L/min in adults to accomplish a complete purge of the extrathoracic anatomic reservoir between breaths.

DETAILED DESCRIPTION:
All patients were submitted to, History, Clinical examination, ABG, Laboratory assessment: as needed, ICU scores: APACHE II score.

Weaning from mechanical ventilation procedure:

The procedure of weaning from mechanical ventilation will be considered as early as possible. Patients who received mechanical ventilation >24 h will receive daily screening of subjective and objective indices for assessment of readiness to wean. Weaning will be conducted according to the statement of the ERS, ATS, ESICM, SCCM and SRLF.

Subjects who fulfill criteria for weaning readiness will be extubated and randomized in a ratio of 1:1:1 to either HVNI or HFNC or Noninvasive ventilation.

Weaning procedure will be considered successful when the spontaneous breathing is sustained for 48 consecutive hours without respiratory distress, with pH>7.35 and PaO2>60 mm Hg in a patient breathing through a mask at FiO2≤0.5.

The weaning outcome is considered a failure when death occurred within 48 hours of extubation. Initiation of mechanical ventilation within 48 hours of liberation from MV will be also considered to be a failure.

ELIGIBILITY:
Inclusion Criteria:

* Adults (≥18 years) intubated for >24 hours due to acute respiratory failure, identified as high-risk for extubation failure AND fulfilling standard readiness-to-wean criteria (e.g., resolution of cause of intubation, adequate gas exchange [P/F ≥150], hemodynamic stability, spontaneous breathing trial [SBT] success)

Exclusion Criteria:

* Patients with central nervous system disorders unrelated to hypercapnic encephalopathy or hypoxemia.
* Patients with post arrest encephalopathy.
* Patient with previous tracheotomy.
* Patients who received noninvasive ventilation without subsequent intubation.
* Patients with end organ failure.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2024-02-01 (Actual); Primary Completion 2025-09-01 (Estimated); Study Completion 2025-10-01 (Estimated)

PRIMARY OUTCOMES:
Successful weaning | 48 hours
  Weaning procedure will be considered successful when the spontaneous breathing is sustained for 48 consecutive hours without respiratory distress, with pH>7.35 and PaO2>60 mm Hg in a patient breathing through a mask at FiO2≤0.5

CONTACTS AND LOCATIONS:
Overall Officials: waleed gamal elddin, ass. prof, Principal Investigator — Assiut University
Locations (1):
- Assiut University hospital, Asyut, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Longhini F, Pisani L, Lungu R, Comellini V, Bruni A, Garofalo E, Laura Vega M, Cammarota G, Nava S, Navalesi P. High-Flow Oxygen Therapy After Noninvasive Ventilation Interruption in Patients Recovering From Hypercapnic Acute Respiratory Failure: A Physiological Crossover Trial. Crit Care Med. 2019 Jun;47(6):e506-e511. doi: 10.1097/CCM.0000000000003740. PMID 30882477
- [Background] Doshi PB, Whittle JS, Dungan G 2nd, Volakis LI, Bublewicz M, Kearney J, Miller TL, Dodge D, Harsch MR, DeBellis R, Chambers KA. The ventilatory effect of high velocity nasal insufflation compared to non-invasive positive-pressure ventilation in the treatment of hypercapneic respiratory failure: A subgroup analysis. Heart Lung. 2020 Sep-Oct;49(5):610-615. doi: 10.1016/j.hrtlng.2020.03.008. Epub 2020 Apr 6. PMID 32273085